CLINICAL TRIAL: NCT03412877
Title: A Phase II Study Using the Administration of Autologous T-Cells Genetically Engineered to Express T-Cell Receptors Reactive Against Neoantigens in Patients With Metastatic Cancer
Brief Title: Administration of Autologous T-Cells Genetically Engineered to Express T-Cell Receptors Reactive Against Neoantigens in People With Metastatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180049; 18-C-0049
Record Dates: First submitted 2018-01-26; First posted 2018-01-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-08-21

CONDITIONS: Endocrine Tumors; Non-Small Cell Lung Cancer; Ovarian Cancer; Breast Cancer; Gastrointestinal/Genitourinary Cancers; Neuroendocrine Tumors; Multiple Myeloma
Keywords: Gene Therapy; Immunotherapy; Cell Therapy; Adoptive Cell Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Breast Neoplasms; Urogenital Neoplasms; Neuroendocrine Tumors; Multiple Myeloma | interventions — Cyclophosphamide; fludarabine; aldesleukin; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/iTCR (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + Individual Patient TCR-Transduced PBL + high- or low-dose aldesleukin
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin; Biological: Individual Patient TCR-Transduced PBL
- 2/iTCR + Pembro (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + Individual Patient TCRTransduced PBL + high- or low-dose aldesleukin + pembrolizumab prior to cell administration and 3 additional doses every 3 weeksfollowing cell infusion
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin; Biological: Individual Patient TCR-Transduced PBL; Drug: Pembrolizumab (KEYTRUDA(R))

INTERVENTIONS:
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day x 2 days IV in 250 mL D5W infused simultaneously with mesna 15 mg/kg/day over 1 hour x 2 days.
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days.
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 10 doses). Patients in Cohort 3 may receive 72,000 IU/kg IV.
Biological: Individual Patient TCR-Transduced PBL — Day 0: Cells will be infused intravenously on the Patient Care Unit over 20-30 minutes (2-4 days after the last dose of fludarabine).
Drug: Pembrolizumab (KEYTRUDA(R)) — Arm 2: Pembrolizumab 2 mg/kg IV over approximately 30 minutes on Days -2, 21, 42, and 63.
  Arms: 2/iTCR + Pembro

SUMMARY:
Background:

A person s tumor is studied for mutations. When cells are found that can attack the mutation in a person s tumor, the genes from those cells are studied to find the parts that make the attack possible. White blood cells are then taken from the person s body, and the gene transfer occurs in a laboratory. A type of virus is used to transfer the genes that make those white blood cells able to attack the mutation in the tumor. The gene transfer therapy is the return of those white blood cells back to the person.

Objective:

To see if gene transfer therapy of white blood cells can shrink tumors.

Eligibility:

People with certain metastatic cancer for which standard treatments have not worked.

Design:

Participants may complete screening under another protocol. Screening includes:

* Getting tumor cells from a previous procedure
* Medical history
* Physical exam
* Scans
* Blood, urine, heart, and lung tests

The study has 8 stages:

1. Screening tests repeated over 1-2 weeks. Participants will have leukapheresis: Blood is removed by a needle in one arm. A machine removes white blood cells. The rest of the blood is returned by a needle in the other arm.
2. Care at home over approximately 12 weeks.
3. Stopping therapy for 4-6 weeks while their cells are changed in a lab.
4. Hospital stay approximately 3-4 weeks for treatment. An IV catheter will be placed in the chest to administer drugs.
5. Patients on Arm 2 of the study will receive the first dose of pembrolizumab while in the hospital. Three additional doses will be given after the cell infusion 3 weeks apart.
6. Receiving changed cells by catheter. Then getting a drug over 1-5 days to help the cells live longer.
7. Recover in the hospital for 1-2 weeks. Participants will get drugs and have blood and urine tests.
8. Participants will take an antibiotic and maybe an antiviral for at least 6 months after treatment. They will have repeat screening tests at visits every few months for the first year, every 6 months for the second year, then as determined.

DETAILED DESCRIPTION:
Background:

* The administration of autologous tumor-infiltrating lymphocytes (TIL) can mediate complete, durable regressions in 20-25% of participants with metastatic melanoma. Recent studies have shown that these TIL predominantly recognize unique mutated neoantigens expressed by the cancer not shared by other melanomas.
* Administration of bulk autologous TIL to participants with a variety of other solid cancers, including cancers of the gastrointestinal tract and genitourinary tract, have little if any therapeutic impact.
* Recent studies in the National Cancer Institute Surgery Branch (NCI-SB) have shown that TIL from non-melanoma solid cancers can also contain T-cells reactive against non-shared unique mutated or oncoviral neoantigens expressed in the cancer. The frequency of these T-cells is very low (often < 0.1%) and it is thus difficult to isolate and grow mutation reactive T-cells to levels required for effective therapy.
* In a single patient with chemo-refractory metastatic cholangiocarcinoma we were able to grow a relatively pure population of neoantigen reactive TIL and administration of these cells mediated a near-complete regression of all metastatic disease now lasting 2.5 years.
* We have developed approaches to identify these rare neoantigen reactive T-cells from common non-melanoma cancers, to isolate their T-cell receptors (TCR), and to genetically engineer autologous peripheral blood lymphocytes (PBL) to express these TCRs with high efficiency. The neoantigen TCR gene-modified cells can recognize and destroy the autologous cancer in vitro.
* In addition to reactivity to neoantigens derived from nonsynonymous mutations, T-cells can recognize human papilloma virus (HPV) epitopes in participants with HPV- induced cancers. The TCR from these reactive cells can be isolated and retrovirally-transduced into autologous PBL with high efficiency.
* With these techniques, we have isolated a number of TCRs selectively recognizing shared mutated oncogenes (e.g., KRAS, TP53) or shared oncoviral proteins (e.g. HPV) in the context of several major histocompatibility complexes (MHC-I and MHC-II).
* This clinical protocol will treat participants with refractory solid cancers using the adoptive transfer of autologous PBL transduced with genes encoding TCRs that recognize unique mutated or oncoviral neoantigens expressed by the cancer.

Objectives:

-Primary objective:

--Determine the rate of objective response (using RECIST v1.1 criteria) of participants with solid cancers who receive pembrolizumab plus autologous PBL (Arm 2) that have been transduced with genes encoding T-cell receptors that recognize mutated or oncoviral neoantigens in the autologous cancer

Eligibility:

-Participants must be/have:

* Age greater than or equal to 18 years and less than or equal to 72 years
* Metastatic solid cancer with at least one lesion that can be measured, that falls into one of five cohorts: (1) gastrointestinal and genitourinary cancers; (2) breast, ovarian, and other solid cancers; (3) non-small cell lung cancer (NSCLC); (4) endocrine tumors including neuroendocrine tumors and, (5) multiple myeloma with solid masses (plasmacytomas).
* Evaluable solid cancer that has recurred following standard chemotherapy or standard systemic therapy
* Normal basic laboratory values
* No allergies or hypersensitivity to high-dose aldesleukin administration
* No concurrent major medical illnesses or any form of immunodeficiency.

Design:

* Participants will have already undergone resection or biopsy to obtain tumor for generation of autologous TIL cultures. This will have been conducted under the NCI-SB cell harvest protocol 03-C-0277 (Cell Harvest and Preparation for Surgery Branch Adoptive Cell Therapy Protocols).
* Exomic sequencing, and often RNA-Seq will be performed to identify the mutations expressed in the patient s cancer. Multiple autologous TIL cultures will be grown and tested for reactivity against mutations from the autologous tumor using assays we have developed that involve the exposure of autologous antigen-presenting cells to long peptides containing the mutation or tandem mini-genes encoding the mutation.
* T-cell cultures with reactivity against mutations will be identified and the individual T- cell receptors that recognize the mutation will be synthesized and used to create a retrovirus for transduction of the TCR into the patient s autologous PBL.
* Participants that present with tumors expressing oncoviral neoantigens will be treated with autologous PBLs retrovirally transduced with TCR(s) targeting the oncoviral neoantigen.
* Participants that present with tumors expressing mutated shared oncogenes (e.g., KRAS, TP53) or oncoviral proteins (e.g., HPV) that also express the appropriate restriction element may be treated with autologous PBLs retrovirally transduced with TCR(s) previously isolated in the Surgery Branch targeting the shared mutated antigen. These participants will be administered a cell infusion product of TCRs targeting mutated shared oncogenes (e.g., KRAS, TP53) or oncoviral proteins (e.g., HPV). Their cell infusion product will not include PBL transduced with unique (i.e., non-shared) TCR(s).
* Participants will be enrolled into one of five cohorts: (1) metastatic gastrointestinal and genitourinary cancers; (2) metastatic breast, ovarian, and other solid cancers; (3) metastatic non-small cell lung cancer (NSCLC); (4) metastatic endocrine tumors including neuroendocrine tumors and; (5) multiple myeloma with solid masses (plasmacytomas). Autologous PBL transduced with TCR(s) targeting neoantigens (mutated shared oncogenes e.g., TP53, KRAS, individual non-synonymous mutations , or oncoviral proteins) will then be expanded to large numbers using our standard rapid expansion protocol.
* Participants enrolled on Arm 1 and Arm 2 will receive a non-myeloablative, lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the infusion of autologous transduced PBL and high-dose aldesleukin. At the discretion of the Principal Investigator (PI), participants enrolled in Cohort 3 (NSCLC) may receive low-dose aldesleukin.
* Participants enrolled on Arm 2 will receive pembrolizumab prior to cell administration and three additional doses every three weeks following the cell infusion. Participants who have experienced major organ toxicity due to previous treatment with pembrolizumab (or equivalent PD-1/PD-L1 blockade) will be enrolled on Arm 1.
* Clinical and immunologic response will be evaluated about 4-6 weeks after cell infusion and periodically thereafter.
* It is anticipated that approximately one participant per month may enroll on the trial for each of the four histologic cohorts for Arm 2. There will be a limit of 15 participants per cohort enrolled on Arm 1 (75 participants for Arm 1), and accrual of up to 4 x 50 = 200 total evaluable participants on Arm 2. It is expected that once full manufacturing capability is reached, the accrual may be completed in approximately 4-5 years. In order to allow for a small number of inevaluable participants, the accrual ceiling will be set to 285.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Metastatic, solid cancer that can be measured, and falls into one of five cohorts: (1) gastrointestinal and genitourinary cancers; (2) breast, ovarian, and other solid cancers; (3) non-small cell lung cancer (NSCLC); (4) endocrine tumors including neuroendocrine tumors and, (5) multiple myeloma that includes measurable solid tumors (plasmacytomas). Participants with multiple myeloma are potentially eligible only if they have measurable multiple myeloma as defined in Section 16.7 after plasmacytoma resection.

Note: NSCLC includes but is not limited to squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinomas.

* Documented diagnosis of cancer.
* Refractory to approved standard systemic therapy. Specifically:

  * Participants with metastatic colorectal cancer must have received oxaliplatin or irinotecan.
  * Participants with breast and ovarian cancer must be refractory to first- line treatment and refractory to or have refused second-line treatments.
  * Participants with NSCLC must have received at least one platinum-based chemotherapy regimen and at least one FDA-approved targeted treatment (when appropriate).
* Participants with endocrine tumors including neuroendocrine tumors must be refractory to first-line therapy (e.g., lanreotide, octreotide) and must be refractory or have refused second-line treatments such as everolimus, sunitinib, or 177 Lu-Dotatate, if indicated.
* Participants with multiple myeloma must have received at least four prior lines of therapy that included at least one exposure to an immunomodulatory drug such as lenalidomide, a proteosome inhibitor, an anti-CD38 antibody treatment, and an autologous stem cell transplant.
* Participants with three (3) or fewer brain metastases that are < 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month after treatment for the participant to be eligible. Participants with surgically resected brain metastases are eligible.
* Age greater than or equal to 18 years and less than or equal to 72 years.
* Clinical performance status of ECOG 0 or 1.
* Participants of both sexes must be willing to practice birth control from the time of enrollment on this study and for and 12 months after the last dose of combined chemotherapy for individuals of child-bearing potential (IOCBP) and four months after treatment for participants who can father a child.
* Individuals of child-bearing potential must be willing to undergo a pregnancy test prior to the start of treatment because of the potentially dangerous effects of the treatment on the fetus.

NOTE: Certain malignancies may secrete hormones that produce false positive pregnancy tests. Serial blood testing (e.g. HCG measurements) and/ or ultrasound may be performed for clarification.

* Serology:

  * Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Participants who are HIV seropositive may have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then participant must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Hematology:

  * ANC > 1000/mm^3 without the support of filgrastim
  * WBC greater than or equal to 2500/mm^3
  * Platelet count greater than or equal to 80,000/mm^3
  * Hemoglobin > 8.0 g/dL. Subjects may be transfused to reach this cut-off.
* Chemistry:

  * Serum ALT/AST less than or equal to 5.0 x ULN
  * Serum creatinine less than or equal to 1.6 mg/dL.
  * Total bilirubin less than or equal to 2.0 mg/dL, except in participants with Gilbert's Syndrome, who must have a total bilirubin less than or equal to 3.0 mg/dL.
* Participants must have completed any prior systemic therapy at the time of enrollment.

Note: Participants may have undergone minor surgical procedures or limited field radiotherapy within the four weeks prior to enrollment, as long as related major organ toxicities have recovered to grade 1 or less. In addition, participants with multiple myeloma may receive bridging therapy during the time between study enrollment and start of study therapy. This may be necessary due to the long time needed for cell production on this study. After bridging therapy and within 14 days of protocol treatment start, participants with multiple myeloma must still have measurable multiple myeloma.

* For Cohort 3: More than two weeks must have elapsed since any prior palliation for major bronchial occlusion or bleeding at the time the patient receives the preparative regimen, and patient s toxicities must have recovered to a grade 1 or less.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Willing to sign a durable power of attorney.
* Subjects must be co-enrolled on protocol 03-C-0277.

EXCLUSION CRITERIA:

* Participants who are pregnant or nursing because of the potentially dangerous effects of the treatment on the fetus or infant.
* Concurrent systemic steroid therapy.
* Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses.
* For Cohort 3: Any major bronchial occlusion or bleeding not amenable to palliation.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS).
* History of major organ autoimmune disease.
* For Arm 2: Grade 3 or 4 major organ irAEs following treatment with anti-PD-1/PD-L1, including but not limited to myocarditis and pneumonitis.

Note: Participants with grade 3 or 4 major organ irAEs may be enrolled on Arm 1 if all other eligibility criteria are met.

* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Participants who have decreased immune-competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
* For Cohorts 1, 2, 4. or 5: Clinically significant participant history which in the judgment of the Principal Investigator (PI) would compromise the participants ability to tolerate high-dose aldesleukin.

Note: At the discretion of the PI, participants enrolled in Cohort 3 may receive low-dose aldesleukin.

* History of coronary revascularization or ischemic symptoms.
* For select participants with a clinical history prompting cardiac evaluation: last known LVEF less than or equal to 45%.
* For select participants with a clinical history prompting pulmonary evaluation: known FEV1 less than or equal to 50% predicted.
* Participants who are receiving any other investigational agents.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2018-09-06 (Actual); Primary Completion 2027-03-23 (Estimated); Study Completion 2028-03-23 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 and 12 weeks after cell infusion, then every 3 months x3, then every 6 months x 2 years, then per PI discretion
  Percentage of patients who receive pembrolizumab as part of the treatment regimen that have a clinical response to treatment (objective tumor regression)

SECONDARY OUTCOMES:
Safety and tolerance | 6 weeks ( 2 weeks) following administration of the cell product or 30 days following the last dose of pembrolizumab
  Using standard CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Tran E, Turcotte S, Gros A, Robbins PF, Lu YC, Dudley ME, Wunderlich JR, Somerville RP, Hogan K, Hinrichs CS, Parkhurst MR, Yang JC, Rosenberg SA. Cancer immunotherapy based on mutation-specific CD4+ T cells in a patient with epithelial cancer. Science. 2014 May 9;344(6184):641-5. doi: 10.1126/science.1251102. PMID 24812403
- [Background] Lu YC, Yao X, Crystal JS, Li YF, El-Gamil M, Gross C, Davis L, Dudley ME, Yang JC, Samuels Y, Rosenberg SA, Robbins PF. Efficient identification of mutated cancer antigens recognized by T cells associated with durable tumor regressions. Clin Cancer Res. 2014 Jul 1;20(13):3401-10. doi: 10.1158/1078-0432.CCR-14-0433. PMID 24987109
- [Background] Robbins PF, Lu YC, El-Gamil M, Li YF, Gross C, Gartner J, Lin JC, Teer JK, Cliften P, Tycksen E, Samuels Y, Rosenberg SA. Mining exomic sequencing data to identify mutated antigens recognized by adoptively transferred tumor-reactive T cells. Nat Med. 2013 Jun;19(6):747-52. doi: 10.1038/nm.3161. Epub 2013 May 5. PMID 23644516
- [Derived] Parkhurst M, Goff SL, Lowery FJ, Beyer RK, Halas H, Robbins PF, Prickett TD, Gartner JJ, Sindiri S, Krishna S, Zacharakis N, Ngo L, Ray S, Bera A, Shepherd R, Levin N, Kim SP, Copeland A, Nah S, Levi S, Parikh N, Kwong MLM, Klemen ND, Yang JC, Rosenberg SA. Adoptive transfer of personalized neoantigen-reactive TCR-transduced T cells in metastatic colorectal cancer: phase 2 trial interim results. Nat Med. 2024 Sep;30(9):2586-2595. doi: 10.1038/s41591-024-03109-0. Epub 2024 Jul 11. PMID 38992129
- [Derived] Levin N, Kim SP, Marquardt CA, Vale NR, Yu Z, Sindiri S, Gartner JJ, Parkhurst M, Krishna S, Lowery FJ, Zacharakis N, Levy L, Prickett TD, Benzine T, Ray S, Masi RV, Gasmi B, Li Y, Islam R, Bera A, Goff SL, Robbins PF, Rosenberg SA. Neoantigen-specific stimulation of tumor-infiltrating lymphocytes enables effective TCR isolation and expansion while preserving stem-like memory phenotypes. J Immunother Cancer. 2024 May 30;12(5):e008645. doi: 10.1136/jitc-2023-008645. PMID 38816232
- [Derived] Kooragayala K, Lou J, Hong YK. Current State of Cell Therapies for Gastrointestinal Cancers. Cancer J. 2022 Jul-Aug 01;28(4):310-321. doi: 10.1097/PPO.0000000000000611. PMID 35880941
- [Derived] Levy PL, Gros A. Fast track to personalized TCR T cell therapies. Cancer Cell. 2022 May 9;40(5):447-449. doi: 10.1016/j.ccell.2022.04.013. Epub 2022 May 9. PMID 35537408
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-C-0049.html